CLINICAL TRIAL: NCT01287871
Title: Addressing Stigma in Screening and Diagnostic Delay for Cervical Cancer
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 09136
Record Dates: First submitted 2011-01-31; First posted 2011-02-02 (Estimated); Last update posted 2025-06-26 (Actual); Status verified 2025-06

CONDITIONS: Cervical Cancer Screening
Keywords: Cervical Cancer Screening
MeSH Terms: interventions — Palliative Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Social media intervention (Other): Women between the ages of 18-70 who have not been diagnosed with any type of cancer and are of African descent or Latina
  Interventions: Other: supportive care

INTERVENTIONS:
Other: supportive care

SUMMARY:
This study aims to 1) implement a culturally and contextually rooted innovative multifoci, social marketing intervention involving societal focused media campaign elements to break down the barriers and facilitate timely and appropriate screening practices for cervical cancer; 2) measure cervical cancer stigma from a culturally relevant theoretical and conceptual framework; and 3) assess the influence of stigma on hindering seeking the PAP test. Further, this is an international study that will bring together a multi-disciplinary investigatory team, community advocates and State health agencies to deliver a social marketing intervention in Southern California (the Inland Empire region specifically) and Trinidad and Tobago.

ELIGIBILITY:
Inclusion Criteria:

Women will be included if they:

1. have not been diagnosed with any type of cancer
2. are between the ages of 18-70
3. self-identify as being African descended or Latina
4. are able to speak English and/or Spanish
5. acknowledge that a Pap test is currently needed

Exclusion Criteria:

1. Cervical cancer is diagnosed only in women, therefore this study only includes women
2. Women who have been and/or are currently diagnosed with any type of cancer will be excluded
3. Women with other major medical conditions (e.g. stroke and degenerative illness) will be excluded
4. During the screening the level of symptomatology for depression and anxiety will be assessed. Women with severe depression and anxiety will be excluded, but appropriate psychological follow-up and referral will be provided
5. Women older than 70 years will be excluded

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 336 (Actual)
Dates: Start 2011-01; Primary Completion 2012-10 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Evaluation of the ability of the social media intervention "End Stigma End Fear, End Cervical Cancer" to counter stigma of cervical cancer among disadvantaged women who acknowledge needing a Pap test at pre-intervention baseline | 3 months after the intervention is implemented
  To evaluate the ability of the social media intervention "End Stigma End Fear, End Cervical Cancer" to counter stigma of cervical cancer, by determining whether, among disadvantaged women who acknowledge needing a Pap test at pre-intervention baseline, degree of exposure to the intervention is associated with the following endpoints at 3 months after the intervention is implemented:
  1. post-intervention change in stigma score relative to pre-intervention, and
  2. Pap testing (scored as 0=made no attempt, 1=made some attempt but did not get tested, 2=obtained Pap test).

SECONDARY OUTCOMES:
Assessment of whether change in stigma score is associated with Pap testing. | 3 months after the intervention is implemented
Identification of factors associated with exposure to the intervention overall and to its individual components | 3 months after the intervention is implemented
Assessment of whether each component of the intervention is associated with the study endpoints, by testing the 4 components (billboards/posters, newspaper advertisements, health brochures, and radio announcements) rather than the overall exposure score | 3 months after the intervention is implemented

CONTACTS AND LOCATIONS:
Overall Officials: Kimlin Ashing-Giwa, PhD, Principal Investigator — City of Hope Medical Center
Locations (1):
- City of Hope Medical Center, Duarte, California, United States